CLINICAL TRIAL: NCT05392907
Title: Forensic-medical Aspects of Lower Limb Prosthetics: An Observational Study
Acronym: CP-PRO-01-20
Status: Completed | Type: Observational
Sponsor: Istituto Nazionale Assicurazione contro gli Infortuni sul Lavoro (Other)
Responsible Party: Sponsor
Other Study IDs: 747-2020-OSS-AUSLBO-20124
Record Dates: First submitted 2022-05-11; First posted 2022-05-26 (Actual); Results first posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-04

CONDITIONS: Amputation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study investigated the perceived-mobility of patients with unilateral lower limb amputations by means of patient-reported outcome measures (PROMs). Such aspect may play an important role in evaluating the patient impairment and addressing forensic-medical issues. However, to this concern, the use of PROMs has not been extensively investigated yet. Among the validated PROMs, the study assessed self-perceived mobility and quality of life by administering the Trinity Amputation Prosthetic Evaluation Survey (TAPES) and the more recent Prosthetic Mobility Questionnaire (PMQ). The aim of this observational study was to improve the estimation of the physical and psychological impairment caused by the amputation, focusing on the impact of the limb loss on social participation, quality of life and daily living activities.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 18 and 65 years
* Unilateral trans-femural or trans-tibial amputation
* Experienced prosthesis users (at least two years)
* Subjects that provided written informed consent to study participation and data publication

Exclusion Criteria:

* Severe comorbidities
* Psychological impairment
* Pregnancy
* Patient not collaborative

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Subjects with a unilateral lower limb amputation either trans-femural or trans-tibial
  * Age:18-65 years old
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2021-07-23 (Actual); Study Completion 2021-07-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Protesi Inail, Budrio, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided
The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request

RESULTS

PARTICIPANT FLOW:
Groups:
- Lower Limb Amputation: Subjects with a unilateral lower limb amputation, even trans-femural or trans-tibial
Period: Overall Study
Arm/Group | Lower Limb Amputation
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lower Limb Amputation
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 50
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 50 [23 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 50
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Italy | 50
Amputation level (trans-femural) [Number; unit: participants] | 25

OUTCOME MEASURES:

1. Primary Outcome: Questionnaire: Trinity Amputation Prosthesis Experience Scale (TAPES)
Description: The questionnaire investigates three aspects of the quality of life of lower limb amputee subjects:
  1. psychosocial adjustment: 15 items, 5-point rating scale, score range: 15-75, higher scores indicates greater levels of adjustment. Therefore, higher values represent a better outcome.
  2. activity restriction: 12 items, 4-point rating scale, score range: 0-24, higher scores indicates greater activity restriction. Therefore, higher values represent a worse outcome.
  3. prosthetic satisfaction: 15 items, 5-point rating scale, score range: 10-50, higher scores indicates greater satisfaction with the prosthesis. Therefore, higher values represent a better outcome.
  Results of psychosocial adjustment, activity restriction, and prosthetic satisfaction are presented separately.
Time Frame: After recruitment, patient anamnesis is performed by an expert clinician. Then, the TAPES questionnaire is administered. The completion time is about 15 minutes
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Lower Limb Amputation: People with unilateral trans-femoral or trans-tibial amputatio
Arm/Group | Lower Limb Amputation
Number analyzed (Participants) | 50
units on a scale
  Psychosocial adjustment | 57 [52 to 63.25]
  Activity restriction | 8 [4.75 to 11]
  Prosthetic satisfaction | 40 [37 to 44.25]

2. Primary Outcome: Score of the Prosthetic Mobility Questionnaire (PMQ)
Description: The "Prosthetic Mobility Questionnaire" (PMQ), available in the Italian version, investigates self-perceived mobility through 12 items. Each item score ranges 0-4 for a total score ranging between 0 and 48. The higher the score, the higher the self-perceived level of mobility.
Time Frame: After completion of TAPES questionnaire, PMQ is administered. The completion time is about 3 minutes.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Lower Limb Amputation
Number analyzed (Participants) | 50
units on a scale | 31.5 [25 to 35]

ADVERSE EVENTS:
Time Frame: 9 months
Description: No adverse events may occur because the objective of the study is exclusively related to questionnaire completion
Arm/Group | Lower Limb Amputation
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-29): https://cdn.clinicaltrials.gov/large-docs/07/NCT05392907/Prot_SAP_000.pdf